CLINICAL TRIAL: NCT06974097
Title: Tumor Associated Neutrophils as a Biomarker of Chemo-immunotherapy Response in Locally Advanced Non-small Cell Lung Cancer : a Model Based on Neoadjuvant Strategy
Acronym: NEO-TAN
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL24_0275
Record Dates: First submitted 2025-05-07; First posted 2025-05-15 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: blood sampling — blood sampling

SUMMARY:
evaluate the predictive value of circulating neutrophil DNA methylation profiles, identified from the ALCINA 2 cohort, on pre-treatment blood samples (T0), for the histological response to neoadjuvant chemo-immunotherapy in patients with resectable non-small cell lung cancer (NSCLC)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Resectable non-small cell lung cancer (NSCLC), stage IIA to IIIB.
* Lymph node status obtained by Positron Emission Tomoscintigraphy (PET)-scanner, confirmation of lymph node status by optional histological sampling (mediastinoscopy, thoracoscopy, echo-endoscopy).
* No secondary lesions in the cerebrum or extra-cerebrum confirmed on brain MRI, PET scanner +/- injected cerebro-thoraco-abdomino-pelvic scanner.
* Neoadjuvant immunochemotherapy strategy validated by a multidisciplinary consultation meeting (RCP) prior to the start of treatment.
* Lung function compatible with thoracic surgery, patient meets surgical and anesthetic criteria for operability
* Measurable disease according to RECIST criteria version 1.1

Exclusion Criteria:

* Previous systemic treatment for the same CBNPC.
* Diagnosis of another solid tumor within the last 3 years, ‡ excluding non melanoma cutaneous and cervical carcinomas .
* Contraindication to immunotherapy.
* Non-objection to participate in research not collected.
* Patients unable to read and/or write.
* Inability to monitor patient during study period
* Persons unable to express their consent.
* Not affiliated to a social security scheme.
* Persons under court protection.
* Persons participating in another research study with an ongoing exclusion period.
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years, older with resectable, locally advanced non-small cell lung cancer (NSCLC) at high risk of recurrence, eligible for neoadjuvant chemo-immunotherapy
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2028-07-28 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Area under the ROC curve (AUC) of neutrophil DNA methylation profiles for predicting histologic response | 6 Months after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Camille TRAVERT, Doctor of Medicine, Principal Investigator — CHU de Montpellier
Locations (1):
- CHU de Montpellier - Hôpital Arnaud de Villeneuve, Montpellier, Cedex 5, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mistry P, Nakabo S, O'Neil L, Goel RR, Jiang K, Carmona-Rivera C, Gupta S, Chan DW, Carlucci PM, Wang X, Naz F, Manna Z, Dey A, Mehta NN, Hasni S, Dell'Orso S, Gutierrez-Cruz G, Sun HW, Kaplan MJ. Transcriptomic, epigenetic, and functional analyses implicate neutrophil diversity in the pathogenesis of systemic lupus erythematosus. Proc Natl Acad Sci U S A. 2019 Dec 10;116(50):25222-25228. doi: 10.1073/pnas.1908576116. Epub 2019 Nov 21. PMID 31754025
- [Background] Engblom C, Pfirschke C, Zilionis R, Da Silva Martins J, Bos SA, Courties G, Rickelt S, Severe N, Baryawno N, Faget J, Savova V, Zemmour D, Kline J, Siwicki M, Garris C, Pucci F, Liao HW, Lin YJ, Newton A, Yaghi OK, Iwamoto Y, Tricot B, Wojtkiewicz GR, Nahrendorf M, Cortez-Retamozo V, Meylan E, Hynes RO, Demay M, Klein A, Bredella MA, Scadden DT, Weissleder R, Pittet MJ. Osteoblasts remotely supply lung tumors with cancer-promoting SiglecFhigh neutrophils. Science. 2017 Dec 1;358(6367):eaal5081. doi: 10.1126/science.aal5081. PMID 29191879
- [Background] Akbay EA, Koyama S, Liu Y, Dries R, Bufe LE, Silkes M, Alam MM, Magee DM, Jones R, Jinushi M, Kulkarni M, Carretero J, Wang X, Warner-Hatten T, Cavanaugh JD, Osa A, Kumanogoh A, Freeman GJ, Awad MM, Christiani DC, Bueno R, Hammerman PS, Dranoff G, Wong KK. Interleukin-17A Promotes Lung Tumor Progression through Neutrophil Attraction to Tumor Sites and Mediating Resistance to PD-1 Blockade. J Thorac Oncol. 2017 Aug;12(8):1268-1279. doi: 10.1016/j.jtho.2017.04.017. Epub 2017 May 6. PMID 28483607
- See also: Related Info — https://www.e-cancer.fr/Professionnels-de-sante/Les-chiffres-du-cancer-en-France/Epidemiologie-des-cancers/Les-cancers-les-plus-frequents/Cancer-du-poumon.
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/30280635/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/32150489/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/33872070/